CLINICAL TRIAL: NCT05696041
Title: Wrist Stabilizing Exercise Versus Hand Orthotic Intervention for Persons With Hypermobility -A Randomized Clinical Trial
Brief Title: Wrist Stabilizing Exercise Versus Hand Orthotic Intervention for Persons With Hypermobility
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Göteborg University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Gothenburg University
Record Dates: First submitted 2023-01-05; First posted 2023-01-25 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Musculoskeletal Diseases; Joint Instability
Keywords: Therapeutics; Rehabilitation; Quality of Life
MeSH Terms: conditions — Musculoskeletal Diseases; Joint Instability

STUDY DESIGN:
Intervention Model Description: A Randomized Clinical Trial
Who Masked: Participant, Care Provider
Masking Description: Subjects were data randomized to the intervention group or control group in the order in which the signed consent forms were received.
  Occupational therapy in the Primary Care received information, training, and a manual with study protocols on procedures and the names of the included subjects, approximately three weeks before the start of studies.
  Neither OTs nor participants knew which intervention the subjects were randomized to until the envelopes were opened.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The exercise group (WSE) (Experimental): Initial static strength training program for the wrist, which could progress to a higher weight in kilos alternatively to a dynamic strength training program
  * Information about HSD/hEDS
  * Daily exercise
  * Training schedule
  * 3-4 return visits to the OT
  Interventions: Other: Static strength training program or/and Dynamic strength training program of the hand
- Conventional intervention (HO) (No Intervention): * Prescribed the wrist´s with plastic or metal orthoses
  * Information about HSD/hEDS
  * Use the orthosis in specific activities; carrying, vacuuming, doing laundry, driving, bicycling
  * Training schedule
  * 3-4 return visits to the OT

INTERVENTIONS:
Other: Static strength training program or/and Dynamic strength training program of the hand — Four of the five exercises included in the static or dynamic training program were based on holding the weight over the edge of the table and maintaining the position for 10 seconds, then resting briefly and changing to the next position. The training was performed in the following assumed positions, pronation, supination, radial and ulnar position. In the fifth and final exercise, you would squeeze an exercise ball as hard as possible without pain. The starting weight was 0.5 kilogram, and each exercise (1-4) was performed in three sets in the first week. The training increased by one set per week for up to eight sets/week if pain or paresthesia got worsened. If the training worked, the OT and the subject could choose to increase the weight to 1 kilogram and start over with three sets/day and gradually increase the training or switch to a dynamic training program.
  Arms: The exercise group (WSE)

SUMMARY:
The goal of this study is to investigate if a Wrist Stabilizing Exercise Programme, WSE, compared to Conventional Intervention use of orthosis in daily activities, HO in persons with Hypermobility Spectrum Disorders, HSD or hypermobility Ehlers Danlos Syndrome, hEDS, in order to reduce pain and or paraesthesia in the hand.

Participants are persons with HSD and hEDS with symptoms of persistent or intermittent pain and or paraesthesia in the hands for the past three years.

The main question aims to answer

* if the WSE has effect on occupational performance and health related quality of life
* if the WSE has effect on handfunction and handstrength The intervention WSE aimed to improve wrist stabilization and increased grip strength according to a training program.

Researchers will compare WSE and HO to see if there were changes between and within the intervention group, WSE and Convention group.

DETAILED DESCRIPTION:
HSD and hEDS involves connective tissue and is characterized by hypermobility, pain and skin manifestations.

It is unknown whether persons with HSD and hEDS suffer from pain and or paraesthesia in the hands, which contributes to impaired hand function and grip strength, and it is unknown how it affects work performance and health-related quality of life. The purpose of the study was to investigate the effect of wrist stabilizing exercises WSE compared to conventional intervention HO, including orthosis, in persons with HSD and hEDS in order to reduce pain and or paraesthesia in the hand. In addition, the study examined how the interventions affected occupational performance and health-related quality of life as well as effects on function and strength.

Method The samples consisted of adults with HSD and hEDS with symptoms of persistent or intermittent pain and or paraesthesia in the hands for the past three years. WSE aimed at better wrist stabilization and increased grip strength according to a training program. The HO groups intervention included a hand orthosis during daily activities. The study examined changes between and within the interventions of WSE and HO over 12 weeks.169 subjects agreed to participate in the study and were randomized to WSE n = 83 or HO n = 86.

Measurements at baseline, after the end of the intervention and after 6 and 12 months.

The intervention WSE consited of Initial static strength training program for the wrist, which could progress to a higher weight in kilos alternatively to a dynamic strength training program. Information about HSD and hEDS. Daily exercise. Training schedule. 3-4 return visits to the OT.

The conventional HO Prescribed the wrist´s with plastic or metal orthoses. Information about HSD and hEDS. Use the orthosis in specific activities; carrying, vacuuming, doing laundry, driving, bicycling. Training schedule. 3-4 return visits to the OT.

Measurement instruments; JAMAR dynamometer, Disability arm, shoulder and hand Dash, Grip Ability Test GAT, EQ5D.

Approximately 20-25 Occupational Terapists OT with experience of hand training attended a half-day training session and were informed about the study design. The OTs were given a manual for conducting the study. The manual contained information on how the study protocol was to be handled and documented and how the information was to be presented to the subjects. The OTs were trained in the use and administration of the assessment instruments.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years and older
* The diagnosis of HSD/hEDS within the last three years, with intermittent or consistent pain, and/or paresthesia of the hand.
* Swedish speaking

Exclusion Criteria:

* Another illness/injury, such as stroke or arm/hand fracture/injury during the past 6 months, combined with HSD/hEDS, which could have affected the study's results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 169 (Actual)
Dates: Start 2014-08-01; Primary Completion 2014-12-31 (Actual); Study Completion 2016-01-31 (Actual)

PRIMARY OUTCOMES:
DASH questionnaire | Baseline 12 weeks 6 and 12 month
  A self-report instrument measuring capacity involving the shoulder arm and hand. The score is from 0-100 with 0 being no incapacities and 100 for the stated A change of more than 10 points on the DASH score as clinically significant.

SECONDARY OUTCOMES:
The EuroQol EQ-5D | Baseline 12 weeks 6 and 12 month
  A self-report measurement for health-related quality of life. The questionnaire consists of ranked increments from 1-3, where the person checks the option that best fits their current state of health. The second part consists score of perceived health status. A visual analogue scale, graded from 0-100.
The Jamar dynamometer | Baseline 12 weeks 6 and 12 month
  Hand strength. Measured by the right and left hand three times. The Norm range score is based on numeric values for age and gender by North Coast TM Hand Dynamometer. Values below the reference values are considered reduced hand strength and values above the reference values are considered better than normal hand strength. The Norm Ranges differ for differing age intervals. Norm Ranges are also different for gender.
The Grip Ability Test | Baseline 12 weeks 6 and 12 month
  Measure the function of the hand consisting of three sub-tasks. The reference value was numerical and had an average value of 16.5. A normal interval is considered between 11-20. Values above 20 indicate impaired hand function and values below 11 are considered above normal.

CONTACTS AND LOCATIONS:
Locations (1):
- Gothenburg University, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No